CLINICAL TRIAL: NCT03514576
Title: Pasireotide in the Treatment of Hypoglycemia Following Gastric Bypass Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Christfort Øhrstrøm, MD, ph.d. student, Zealand University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PasHypo
Record Dates: First submitted 2018-04-19; First posted 2018-05-02 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Hypoglycemia, Reactive
Keywords: gastric bypass; hypoglycemia; hyperinsulinemia
MeSH Terms: conditions — Hypoglycemia; Hyperinsulinism | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pasireotide75 (Experimental): 75 micrograms Pasireotide 0.3 MG/ML s.c. before a meal tolerance test (MTT)
  Interventions: Drug: Pasireotide 0.3 MG/ML; Diagnostic Test: Meal tolerance test (MTT)
- Pasireotide150 (Experimental): 150 micrograms Pasireotide 0.3 MG/ML s.c. before a meal tolerance test (MTT)
  Interventions: Drug: Pasireotide 0.3 MG/ML; Diagnostic Test: Meal tolerance test (MTT)

INTERVENTIONS:
Drug: Pasireotide 0.3 MG/ML — See arm description
  Other Names: Signifor
Diagnostic Test: Meal tolerance test (MTT) — Subjects will consume the liquid meal at baseline and blood will be drawn for continuous blood sampling.

SUMMARY:
Postprandial hyperinsulinemic hypoglycemia is a well-known and potentially severe complication of Roux-en-Y gastric bypass (RYGB), and the treatment options are limited. Pasireotide has shown to be effective in preventing hypoglycemia in RYGB operated subjects, however treatment often leads to increased hyperglycemia.

The purpose of this study is to investigate two doses of pasireotide that are lower than doses previously used in RYGB operated subjects with postprandial hyperinsulinemic hypoglycemia.

DETAILED DESCRIPTION:
With the growing number of RYGB operated subjects the attention on complications such as postprandial hyperinsulinemic hypoglycemia (PHH) has increased. PHH is characterized by increased glycemic variability and hypoglycemic episodes occurring 2-3 hours after a meal together with a markedly increase in insulin and glucagon-like-peptide 1 (GLP-1) levels. Symptoms vary from dizziness and palpitations to confusion, loss of consciousness and convulsions. At present there are few treatment options available for RYGB patients with PHH and most of them rely on dietary changes that are difficult to adhere to.

Pasireotide has been shown to reduce hypoglycemia in RYGB operated subjects with PHH, but often leads to increased hyperglycemia as well.

The purpose of the study is to investigate two doses of pasireotide in RYGB operated subjects with PHH.

Each subject will undergo two meal tolerance test (MTT) preceded by either 75 µg or 150 µg of pasireotide. Blood samples will be collected throughout the meal test at predefined time points and will be analyzed for glucose, insulin, C-peptide, GLP-1 and glucagon levels.

ELIGIBILITY:
Inclusion Criteria:

* RYGB operated patients with documented hypoglycemia (blood glucose <3.9 mmol/L) who have previously completed the study 'Treatment of hypoglycemia following gastric bypass surgery' (HypoGB2015)
* Hemoglobin > 7,3 mmol/L
* Negative human chorionic gonadotropin (hCG) urine test
* Females of reproductive age: use of safe contraception

Exclusion Criteria:

* Treatment for cardiovascular disease
* Treatment with antipsychotic medication
* Treatment for thyroid disease
* Prior medical treatment of postprandial hyperinsulinemic hypoglycemia
* Prior allergic reactions to the study medicine

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in glucose (mmol/L) in response to a meal tolerance test (MTT) | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes in incremental area under the curve (iAUC) for glucose, nadir glucose values, peak glucose values, time spent with glucose values in the hyperglycemic (>7.8 mmol/L) and the hypoglycemic (<3.9 mmol/L) range

SECONDARY OUTCOMES:
Heart rate | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes heart rate (beats/min) during the course of a meal tolerance test (MTT)
Serum insulin levels | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes in insulin (pmol/L) in response to a meal tolerance test (MTT)
Serum C-peptide levels | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes in C-peptide (nmol/L) in response to a meal tolerance test (MTT)
Plasma glucagon levels | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes in glucagon (pmol/L) in response to a meal tolerance test (MTT)
Plasma GLP-1 levels | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes in glucagon-like peptide 1 (pmol/L) in response to a meal tolerance test (MTT)
Blood pressure | From 20 minutes prior to a liquid test meal to 180 minutes following the meal ingestion
  Changes in blood pressure (mmHg) in response to a meal tolerance test (MTT)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline C Øhrstrøm, MD, Principal Investigator — Department of Medicine, Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No